CLINICAL TRIAL: NCT03189251
Title: Moderate Intake of High Fructose Corn Syrup Sweetened Soft Drinks, Fruit Drinks and Apple Juice Increases Asthma Risk - the Framingham Offspring Cohort
Brief Title: HFCS, Apple Juice, Excess Free Fructose & asthma-the FHS-OS
Status: Completed | Type: Observational
Sponsor: Luanne R DeChristopher (Individual)
Collaborators: Jaime Uribarri, M.D. (Unknown); Katherine L. Tucker, Ph.D. (Unknown)
Responsible Party: Sponsor-Investigator, Luanne R DeChristopher, Independent Researcher, DeChristopher, Luanne R.
Organization: DeChristopher, Luanne R. (Individual)
Other Study IDs: EFF, HFCS, asthma-the FHS-OS
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Eating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dietary intakes — Analysis of association between consumption of high excess free fructose (EFF) beverages (high fructose corn syrup sweetened soft drinks, fruit drinks, apple juice)

SUMMARY:
Perform an exploratory analysis of association between consumption of high excess free fructose (EFF) beverages (high fructose corn syrup sweetened soft drinks, fruit drinks, apple juice) and Chronic Bronchitis (CB)/history of CB, and asthma/ history of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the FHS Offspring who answered questions in the FFQ about soft drinks, fruit drinks and fruit juice consumption; Participants with non-missing data for the exposures and potentially confounding variables of interest.

Exclusion Criteria:

* Extreme energy intake on food frequency questionnaire (defined as ≤600 kcal/day or ≥4800 kcal/day)

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the Framingham Heart Study (Offspring) cohort
Sampling Method: Non-Probability Sample
Enrollment: 2657 (Actual)
Dates: Start 1971-06 (Actual); Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Asthma | Exams 3 - 7, 17 years of follow-up
  Incident asthma defined as self-reported asthma (at each exam), including wheezing or asthma (have you had asthma/ wheeze since the last exam of short duration, long duration or with respiratory infections)

IPD SHARING:
Plan to Share IPD: No